CLINICAL TRIAL: NCT01246401
Title: Naltrexone for Opioid Dependent Released Human Immunodeficiency Virus Positive (HIV+) Criminal Justice Populations
Acronym: NewHope
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Baystate Medical Center (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1007007169; 1K02DA032322-01 (NIH)
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Results first posted 2017-07-17 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2017-06

CONDITIONS: HIV; AIDS; Opioid Dependence; Drug Dependence
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Opioid-Related Disorders; Substance-Related Disorders | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Extended-Release Naltrexone (Active Comparator): Participants will receive intramuscular (IM) injections of Naltrexone once monthly for 6 months, the first injection being prior release
  Interventions: Drug: Extended-Release Naltrexone
- Placebo (Placebo Comparator): Participants will receive IM injections of Placebo once monthly for 6 months, the first injection being prior release
  Interventions: Drug: Extended-Release Naltrexone

INTERVENTIONS:
Drug: Extended-Release Naltrexone — Extended-Release Naltrexone (Vivitrol), once a month by IM injection, for a total of 6 months. Dosage is 380mg
  Other Names: Naltrexone, depot; Vivitrol

SUMMARY:
Specific Aim: To conduct a randomized, placebo-controlled trial of extended release-naltrexone (XR-NTX) among Human Immunodeficiency Virus (HIV) infected prisoners meeting Diagnostic Statistical Manual IV (DSM-IV) criteria for opioid dependence who are transitioning from the structure of a correctional setting to the community.

Hypotheses:

i. XR-NTX will result in improved HIV clinical outcomes, including lower changes in HIV-1 RNA levels, higher CD4 counts and higher rates of retention in care.

ii. XR-NTX will result in improved opioid treatment outcomes, including longer time to opioid relapse, lower addiction severity and lower craving for opioid.

iii. XR-NTX will result in reduced drug- and sex-related HIV risk behaviors compared to the control group.

iv. XR-NTX will result in decreased rates of reincarceration after 12 months of release to the community.

DETAILED DESCRIPTION:
The specific aim for this study is to conduct a placebo-controlled trail (RCT) of XR-NTX among HIV+ persons in jails and prisons meeting DSM-IV criteria for opioid dependence who are transitioning to the community. HIV treatment outcomes (HIV-1 RNA levels, CD4 count, Highly Active Antiretroviral Therapy (HAART) adherence, retention in care), substance abuse (time to relapse to opioid use, % opioid negative urines, opioid craving), adverse side effects and HIV risk behavior (sexual and drug-related risks) outcomes will be compared in 150 recruited prisoners and jail detainees in Connecticut (CT) and Massachusetts (MA) who will be randomized 2:1 to either XR-NTX or placebo. The primary outcome of interest will be the proportion with a HIV-RNA <400 copies/mL at 6 months. Secondary outcomes include mean CD4 count, antiretroviral adherence, retention on HAART and in HIV care, HIV risk behaviors, time-to-relapse to opioid use, percent opioid negative urines, retention on d-NTX and HIV quality of life. Primary and secondary outcomes will be assessed for an additional 6 months after completion of the intervention. If this placebo-controlled trial of XR-NTX among released HIV+ criminal justice system (CJS) persons with opioid dependence demonstrates efficacy and safety, it is likely to become an evidence-based intervention to intervene with this extremely marginalized population in a way that will meet Healthy People 2010's goals to increase the quality and years of life, decrease health disparities particularly among minorities, break the cycle of addiction, reduce the numbers of people within the CJS and launch a number of new and innovative trials and second generation questions for future research. As such, the individual, our health care system and society have a high likelihood to benefit. This will not only be true for strategies here in the U.S., but may have even greater application for geographic areas where the interface between opioid disorders and HIV is even greater.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV criteria for opioid dependence
2. Age > 18 years
3. Confirmed HIV infection, either through positive HIV antibody or detectable HIV-1 RNA level.
4. Within the Connecticut Department of Corrections (CTDOC) or Hampden County Correctional Center (HCCC) and within 30 days of being released to the greater New Haven, Hartford or Springfield areas or within 30 days after release from CTDOC or HCCC.
5. No participation in pharmacotherapy trial in the previous 30 days
6. Not pregnant

Exclusion Criteria:

1. Unable to provide informed consent
2. Verbally or physically threatening to research staff
3. Unable to communicate in either English or Spanish
4. Pending trials for a felony
5. Liver failure (Childs-Pugh Class B or C Cirrhosis)
6. Grade IV Hepatitis (liver function tests > 10X normal)
7. Receiving opioid prescription narcotics or has pain syndrome necessitating future use of opioid prescription narcotics.
8. Receiving active methadone or buprenorphine/naloxone for the treatment of opioid dependency
9. Active opioid withdrawal (within 3-5 days since last opioid ingestion)
10. Pregnancy or unwilling to take contraceptives measures
11. Breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-03; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra A Springer, MD, Principal Investigator — Yale University; Frederick L Altice, Principal Investigator — Yale University
Locations (3):
- United States (3):
  - Yale University, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Baystate Medical Center, Springfield, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
Data has been shared with the National Institute on Drug Abuse as a site in the data harmonization project associated with Seek, Test, Treat and Retain for Criminal Justice Populations.

REFERENCES:
- [Background] Di Paola A, Lincoln T, Skiest DJ, Desabrais M, Altice FL, Springer SA. Design and methods of a double blind randomized placebo-controlled trial of extended-release naltrexone for HIV-infected, opioid dependent prisoners and jail detainees who are transitioning to the community. Contemp Clin Trials. 2014 Nov;39(2):256-68. doi: 10.1016/j.cct.2014.09.002. Epub 2014 Sep 18. PMID 25240704
- [Result] Vagenas P, Di Paola A, Herme M, Lincoln T, Skiest DJ, Altice FL, Springer SA. An evaluation of hepatic enzyme elevations among HIV-infected released prisoners enrolled in two randomized placebo-controlled trials of extended release naltrexone. J Subst Abuse Treat. 2014 Jul;47(1):35-40. doi: 10.1016/j.jsat.2014.02.008. Epub 2014 Mar 12. PMID 24674234
- [Result] Springer SA, Brown SE, Di Paola A, Altice FL. Correlates of retention on extended-release naltrexone among persons living with HIV infection transitioning to the community from the criminal justice system. Drug Alcohol Depend. 2015 Dec 1;157:158-65. doi: 10.1016/j.drugalcdep.2015.10.023. Epub 2015 Oct 28. PMID 26560326
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086
- [Derived] Springer SA, Di Paola A, Azar MM, Barbour R, Biondi BE, Desabrais M, Lincoln T, Skiest DJ, Altice FL. Extended-Release Naltrexone Improves Viral Suppression Among Incarcerated Persons Living With HIV With Opioid Use Disorders Transitioning to the Community: Results of a Double-Blind, Placebo-Controlled Randomized Trial. J Acquir Immune Defic Syndr. 2018 May 1;78(1):43-53. doi: 10.1097/QAI.0000000000001634. PMID 29373393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 151 subjects consented, 58 lost before randomization
Period: Overall Study
Arm/Group | Extended-Release Naltrexone | Placebo
Started | 66 | 27
Completed | 66 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Extended-Release Naltrexone | Placebo | Total
Number analyzed (Participants) | 66 | 27 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (8.3) | 43.9 (7.8) | 45.8 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 55 | 21 | 76
Housing status [Count of Participants; unit: Participants]
  Stable | 23 | 11 | 34
  Unstable | 19 | 4 | 23
  Homeless | 24 | 12 | 36
Currently prescribed ART [Count of Participants; unit: Participants] | 58 | 24 | 82
Alcohol Use Severity (AUDIT score) [Count of Participants; unit: Participants]
  Abstinent or Low-Risk Drinking | 42 | 23 | 65
  Hazardous Drinking | 11 | 2 | 13
  Harmful Drinking | 2 | 0 | 2
  Possible Dependence | 10 | 2 | 12
  Missing | 1 | 0 | 1
Opioid craving [Mean (Standard Deviation); unit: units on a scale] — Opioid craving scale: a 10 item likert scale from 0 to 10 with 10 being highest craving for opioids and 0 representing no craving. Mean scores taken for each group.
  units on a scale | 3.2 (3.6) | 3.5 (3.8) | 3.3 (3.6)
Years Reported use of substances [Mean (Standard Deviation); unit: years]
  Alcohol | 13.5 (15.2) | 9.2 (11.6) | 12.2 (14.3)
  Cannabis | 14 (14.3) | 12.8 (12.5) | 13.6 (13.7)
  Cocaine | 17.5 (11.4) | 18.7 (8.6) | 17.9 (10.6)
  Heroin | 20.1 (11.2) | 18.4 (10.2) | 19.6 (10.9)
  Other Opioids | 2.8 (7.2) | 3.2 (5.4) | 2.9 (6.7)

OUTCOME MEASURES:

1. Primary Outcome: Participants Who Had Undetectable HIV-1 RNA Levels at Less Than 400 Copies/mL at Six Month
Description: Baseline labs will be drawn while subject is in prison, one to three months prior to release. Additionally, labs will be drawn every 3 months for 1 year to monitor changes in HIV-1 RNA levels. Treatment time period was the first 6 months where the primary outcome data will be based on.
Time Frame: 6 months
Population: A total of 80 participants had viral load data at 6 months (56 in XR-NTX group and 24 in Placebo group). The remaining 13 participants (10 in XR-NTX group and 3 in Placebo group) with missing viral load data at 6 months were considered as failure - meaning - having a viral load of 400 or more. Thus included into the final analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 66 | 27
Participants | 45 | 16
Statistical Analysis 1: Comparison: Extended-Release Naltrexone vs Placebo; Test type: Superiority; p = 0.431, Welch's T Test

2. Secondary Outcome: Particpants Who Had Undetectable HIV-1 RNA Levels at Less Than 50 Copies/mL
Description: as for outcome 1
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 66 | 27
Participants | 40 | 11
Statistical Analysis 1: Comparison: Extended-Release Naltrexone vs Placebo; Test type: Superiority; p = 0.087, Welch's T Test

3. Secondary Outcome: CD4 Cell Count (Cells/mL)
Description: Baseline labs will be drawn while subject is in prison, one to three months prior to release. Additional labs will be drawn every 3 months for 1 year to monitor changes in CD4 levels.
Time Frame: Baseline and 6 months
Population: Data was collected via labs. At month 6, due to attrition, data was only available for a total of 46 subjects. These include, 14 in Placebo and 32 in Extended-Release Naltrexone. The mean and STD are presented below.
Measure: Mean (Standard Deviation); unit: cells/ml
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 66 | 27
cells/ml
  Baseline mean CD4 count | 465.2 (273.8) | 580.8 (336.8)
  Month 6 mean CD4 count: number analyzed (Participants) | 32 | 14
  Month 6 mean CD4 count | 462 (306.6) | 485.6 (257.3)

4. Secondary Outcome: Time to Opioid Relapse or End of Intervention
Description: Measuring days to first relapse based on self reported opioids (heroin) use within the 6 month (180 days) intervention period. If participants had no follow-up visits, and thus no self reported opiate use, they were treated as missing. Those who did not relapse within the 6 month intervention period were treated as having 180 days until relapse.
Time Frame: 6 months
Population: Data collected via Time Line Fall Back (TLFB). 15 in XR-NTX group and 4 in Placebo did not have data because of attrition - treated as missing. An additional 19 people in the treatment arm and 9 in placebo filled out the TLFB at 9 or 12 months, and this data was used to fill in missing information.
Measure: Median (Full Range); unit: days
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 51 | 23
days | 137 [0 to 168] | 29 [0 to 168]
Statistical Analysis 1: Comparison: Extended-Release Naltrexone vs Placebo; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney) — Wilcoxon one sided

5. Secondary Outcome: Addiction Severity
Description: The Addiction Severity Index (ASI) questionnaire will be used to assess addiction severity. The ASI composite scoreprovides reliable and valid measure of patient status in a particular module of interest which can then be usecompared at the beginning of treatment to the evaluation endpoint to note the improvement or lack thereof. In this assessment the drug composite score was calculated using algorithm by Treatment Research Institute. If the score increases then it shows increase in severity where as if it decreases then it shows decrease in severity for that measured module. The scale ranges from 0 to 1.
  The mean composite scores for drug use from baseline to 6 months were compared using Nonparametric test.
Time Frame: baseline, and 6 months
Population: An additional subject's data from the experimental group was not collected at baseline. For the 6 months data, the total number of participants with completed assessment used for the analysis was 46 (31 in XR-NTX group and 15 in Placebo group).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 65 | 27
units on a scale
  baseline | 0.37 (0.16) | 0.42 (0.14)
  6 month: number analyzed (Participants) | 31 | 15
  6 month | 0.12 (0.13) | 0.16 (0.16)

6. Secondary Outcome: Craving for Opioids
Description: Craving at baseline compared to 6 month. This is assessed through a self report scale rated 0 to 10; 0 meaning not craving and 10 meaning highest craving. Change in craving score was categorized as 1)no change between baseline and 6 month; 2)increased craving - baseline craving was reported lower than at 6 month; 3)decreased craving - baseline craving was reported higher than 6 month craving.
Time Frame: 6 months
Population: Data available at 6 month determined who was included into the analysis. In this case a total of 47 data points (those with both baseline and 6 month data points) were included into the analysis (32 Extended-Release Naltrexone and 15 Placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 32 | 15
Participants
  No change | 12 | 7
  Increased craving at 6 mo | 6 | 3
  Decreased craving at 6 mo | 14 | 5

7. Secondary Outcome: Antiretroviral Therapy (ART) Adherence 100%
Description: Number of subjects with 100% adherence at 6 months measured using Visual Analogue Scale: 0% to 100%
Time Frame: 6 months
Population: 56 participants with missing data were considered as failure - meaning - with adherence less than 100%, and included into the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 66 | 27
Participants | 25 | 12

8. Secondary Outcome: Participants With Opiate Abstinence Via By Doing Urine Toxicology Test
Description: Percent of subjects with no opiate use at 6 month. Missing data was treated as failure (opiate positive).
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Extended-Release Naltrexone | Placebo
Number analyzed (Participants) | 66 | 27
Participants
  NEG Opi at Day of Release | 44 | 17
  NEG Opi at 6 month | 13 | 5

9. Secondary Outcome: Opioid Abstinence at 6 Months for Those With More Than 4 Injections
Description: Based on self reported opioids (heroin) use. All participants receiving Placebo as well as participants who received 3 or less XR-NTX injections were compared to those who receive 4 or more XR-NTX injection.
Time Frame: 6 months
Population: Collected via Time Line Fall Back (TLFB). Total N analyzed is 74. 12 of the clients had initial or some TLFB data indicating relapse but were counted as lost at 6 months for outcome 4. 19 Clients did not have TLFB data or if they did within 6 month it did not indicate any relapse. These were treated as missing and not included in analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo + Participants With 3 or Fewer XR-NTX Injections: All participants receiving Placebo as well as participants who received 3 or less XR-NTX injections
- 4 or More XR-NTX Injections: All participants who received 4 or more XR-NTX injections
Arm/Group | Placebo + Participants With 3 or Fewer XR-NTX Injections | 4 or More XR-NTX Injections
Number analyzed (Participants) | 58 | 16
Participants | 18 | 13
Statistical Analysis 1: Comparison: Placebo + Participants With 3 or Fewer XR-NTX Injections vs 4 or More XR-NTX Injections; Test type: Superiority; p = 0.03962, Chi-squared

10. Secondary Outcome: ART Adherence for 4 or More Injections XR-NTX Versus Placebo and 3 or Less Injections of XR-NTX
Description: The arm/group number of the participants vary from the primary outcome because this is a treatment effect analysis. All client with missing data at 6 months were considered as failure - meaning - they had less than 100% ART adherence.
Time Frame: 6 months
Population: All client with missing data at 6 months were considered as failure - meaning - they had less than 100% ART adherence.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + Participants With 3 or Fewer XR-NTX Injections | 4 or More XR-NTX Injections
Number analyzed (Participants) | 77 | 16
Participants | 23 | 14

ADVERSE EVENTS:
Arm/Group | Extended-Release Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/27
Other Adverse Events (participants affected / at risk) | 13/66 | 4/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Extended-Release Naltrexone (N=66) | Placebo (N=27)
Headache (Nervous system disorders) | 5 | 0
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 0
Decreased Apetite (Metabolism and nutrition disorders) | 2 | 1
Increased Apetite (Metabolism and nutrition disorders) | 2 | 1
Fatigue (General disorders) | 6 | 1
Skin and Soft Tissue Infection (Skin and subcutaneous tissue disorders) | 2 | 1
Signs of Edema (Blood and lymphatic system disorders) | 2 | 2
Immediate Injection Reaction (Musculoskeletal and connective tissue disorders) | 10 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes